CLINICAL TRIAL: NCT01060839
Title: Evaluation of Partner Notification for Sexually Transmitted Infections in Bangladesh
Brief Title: Evaluation of Counseling for Partner Notification
Acronym: PN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Nazmul Alam, Senior Research Investigator, International Centre for Diarrhoeal Disease Research, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-001; BC#03111459 (Other: ICDDR,B)
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Sexually Transmitted Infections
Keywords: counseling
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single session counseling (Experimental)
  Interventions: Behavioral: Single session counseling
- Standard of care (No Intervention)

INTERVENTIONS:
Behavioral: Single session counseling — For index cases assigned to the counselling arm, a same sex counselor conducted 10-15 minutes individualized sessions. Counselors were specifically trained to deliver partner referral counselling focusing on five issues related to STI prevention and transmission: (1) risk of re-infection if partners are not treated concurrently; (2) risk of developing complications; (3) risk of further spread of infection in the community; (4) the asymptomatic nature of infection; and (5) social obligations and personal coping with an STI.
  Other Names: counseling
  Arms: Single session counseling

SUMMARY:
* In the formative stage of the project, we have investigated through qualitative and quantitative studies to identify a potential intervention to promote partner referral for sexually transmitted patients in Bangladesh.
* We conducted a quasi-randomised trial to evaluate if single session counseling is effective in improving partner referral for patients with sexually transmitted infection.

DETAILED DESCRIPTION:
The study was a quasi-randomized trial, alternating partner referral counselling and standard of care approach for each subsequent patient. First patients was randomly assigned by the project research physician in each clinic then alternative patients allocation was maintained by the study interviewers assigned in each clinic. For index cases assigned to the counselling arm, a same sex counselor conducted 10-15 minutes individualized sessions. Counselors were specifically trained to deliver partner referral counselling focusing on five issues related to STI prevention and transmission: (1) risk of re-infection if partners are not treated concurrently; (2) risk of developing complications; (3) risk of further spread of infection in the community; (4) the asymptomatic nature of infection; and (5) social obligations and personal coping with an STI. Patients in the standard care group received the existing services in the respective clinics, which included clinical consultation, prescription for medication but there was no partner referral counselling per se. In the public clinics, both the counselling and non-counselling group of clients received free medications, while in the NGO clinics they received subsidized fee medications. Both groups also received standard, pre-tested anonymous partner referral cards along with a short briefing by the interviewers that index clients need to hand over this card to their partner(s) to bring them to the respective clinics for assessment of STI status. Partner referral cards were used to follow-up partner referral by tracking the patient identification number and disease code of cards provided by referred patients. In addition, referral cards were useful for the partners to locate the study clinic, to be entitled to free or subsidized medication, and to distinguish the partners from index cases coming to the clinics.

ELIGIBILITY:
Inclusion Criteria:

* Each newly diagnosed STI patients
* Age > 18 years
* Who had a sexual exposure in last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1339 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Proportion of index cases, who referred one or more partner/s to the study clinics within one month of interview. | within one month of interview

CONTACTS AND LOCATIONS:
Overall Officials: Nazmul Alam, DrPH, Principal Investigator — International Centre for Diarrhoeal Disease Resaerch, Bangladesh
Locations (1):
- Dhaka Medical College Hospital, Skin VD out patient clinic, Dhaka, Dhaka Division, Bangladesh